CLINICAL TRIAL: NCT01345565
Title: Hepatocyte Transplantation for Acute Decompensated Liver Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: A funding mechanism is not identified at this time
Sponsor: Ira Fox (Other)
Responsible Party: Sponsor-Investigator, Ira Fox, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO09020051
Record Dates: First submitted 2011-04-26; First posted 2011-05-02 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Liver Failure Acute
Keywords: fulminant hepatic failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — NOS2 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hepatocyte Transplantation (Experimental): See Below
  Interventions: Drug: human hepatocytes

INTERVENTIONS:
Drug: human hepatocytes — The intrahepatic site for liver cell transplantation has been associated with the best engraftment and function based on animal experiments. Several approaches for access to the portal vein will be considered. The technique used will be determined based on what is considered best for the child based on risk/benefit at the time.
  We propose to attempt to infuse approximately 5-10% of the hepatic mass in order to provide improved hepatic function. Since we do not yet know from our experience so far the correct number of cells to transplant in order to improve function, we will continue to infuse hepatocytes as donors become available until the patient improves to the point where they are no longer meet the criteria for organ transplantation. The subject will be evaluated de novo and if they are a candidate for orthotopic liver transplantation they will receive the transplant.

SUMMARY:
The purpose of this research study is to determine whether liver cell transplantation can provide help for patients with liver failure who are unlikely to survive without some form of liver support. The goal of this research study is to determine if liver cell transplants can be effective until a liver transplant is received or until patients recover from their liver failure.

DETAILED DESCRIPTION:
Orthotopic liver transplantation has become the treatment of choice for patients with acute liver failure with poor prognostic signs. Survival following hepatic transplantation has improved in the last decade for a number of reasons. These include improvement in immunosuppression, improved methods for preserving and transporting organs, use of donors which had been previously considered unacceptable, use of reduced-sized grafts , and the use of living-donor hepatic transplantation. Despite encouraging survival statistics, there continues to be significant morbidity and mortality associated with hepatic transplantation. In addition, the success of hepatic transplantation has broadened the indications for this form of therapy without a concomitant increase in the number of donors available for these patients.

Since the development of a method for isolating primary hepatocytes by collagenase perfusion, many investigators have demonstrated the efficacy of hepatocyte transplantation in the treatment of liver failure and inherited metabolic disorders in experimental animals. Treatment of liver diseases with transplantation of isolated hepatocytes rather than the whole liver has several theoretical advantages. Unlike the whole liver, isolated hepatocytes could be cryopreserved for instant availability and could be modified genetically or otherwise to enhance specific functions, stimulate proliferation or abrogate allograft rejection. Hepatocyte transplantation should be less stressful than whole liver transplantation because the host organ remains intact. Since the transplanted cells integrate into the host liver, they could provide restorative potential and the consequences of graft loss would be relatively minor. In addition, hepatocyte transplantation would not interfere with subsequent liver transplantation, should that become necessary.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include those patients with ALF who are potential conventional liver transplant recipient candidates based on PELD criteria as well as those who would not be considered candidates for orthotopic liver transplantation (e.g. patients who appear to be too small or too ill for solid organ transplant or those who have a diagnosis that is a contradiction for whole organ transplantation, for example, systemic mitochondrial hepatopathy).
* If the patient is a candidate for orthotopic liver transplantation (per standard clinical criteria), they will be officially listed for liver transplantation as well as hepatocyte transplantation.
* If a subject is a potential conventional liver transplant recipient candidate and a donor liver is available; the patient will receive a solid organ transplant.
* Subjects ages 0-21 years old will be included in this study.

Exclusion Criteria:

The patient has:

1. Severe cardiovascular or respiratory disease at baseline and at the time of hepatocyte transplant as defined by

   1. Central venous pressure >25 mm Hg or if known, pulmonary capillary wedge pressure of >30 mg Hg or
   2. Oxygen saturation of <90% on > 60% oxygen OR a P/F ratio (Po2/FiO2) of <1.
2. Hemodynamically significant gastrointestinal bleeding causing a systolic blood pressure <70mmHg at the time of transplantation.
3. Uncorrectable coagulopathy despite use of plasmapheresis that would preclude any invasive procedures.
4. Leukopenia at the time of cell transplant, defined as an absolute neutrophil count of <500/µL.
5. Known allergy to immunosuppression medications that are required post transplant procedure for the prevention of rejection.
6. Active malignancy except those with acute liver failure during treatment with estimated life expectancies of >1 year if the malignancy is controlled.
7. Sepsis or other active infection except those without evidence of hemodynamically significant uncontrollable systemic sepsis with positive blood or tissue cultures.
8. Intrauterine pregnancy. All females of childbearing potential will receive a pregnancy test prior to enrollment.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Improvement in evidence of liver function at two weeks after hepatocyte transplant | Two weeks after hepatocyte transplant
  The extent to which hepatocyte transplantation can elicit evidence of improvement in liver function in patients with acute decompensated liver failure not responding to medical management.

SECONDARY OUTCOMES:
Immune Response | two weeks after hepatocyte transplant and monthly thereafter post hepatocyte transplant
  The extent to which the standard immune suppression medications used for solid organ transplantation can effectively control rejection and preserve the function of transplanted hepatocytes without leading to overwhelming infection or other medication related toxicities in the face of hepatic failure.
Quality and Quantity of Hepatocytes | Two weeks after hepatocyte transplant
  The relationship between number and quality of donor hepatocytes infused and engraftment in the livers of patients with the acute liver injury.

CONTACTS AND LOCATIONS:
Overall Officials: Ira J Fox, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fox IJ, Chowdhury JR, Kaufman SS, Goertzen TC, Chowdhury NR, Warkentin PI, Dorko K, Sauter BV, Strom SC. Treatment of the Crigler-Najjar syndrome type I with hepatocyte transplantation. N Engl J Med. 1998 May 14;338(20):1422-6. doi: 10.1056/NEJM199805143382004. No abstract available. PMID 9580649
- [Background] Roger V, Balladur P, Honiger J, Baudrimont M, Delelo R, Robert A, Calmus Y, Capeau J, Nordlinger B. Internal bioartificial liver with xenogeneic hepatocytes prevents death from acute liver failure: an experimental study. Ann Surg. 1998 Jul;228(1):1-7. doi: 10.1097/00000658-199807000-00001. PMID 9671059
- [Background] Habibullah CM, Syed IH, Qamar A, Taher-Uz Z. Human fetal hepatocyte transplantation in patients with fulminant hepatic failure. Transplantation. 1994 Oct 27;58(8):951-2. doi: 10.1097/00007890-199410270-00016. No abstract available. PMID 7940741
- [Background] Gupta S, Aragona E, Vemuru RP, Bhargava KK, Burk RD, Chowdhury JR. Permanent engraftment and function of hepatocytes delivered to the liver: implications for gene therapy and liver repopulation. Hepatology. 1991 Jul;14(1):144-9. doi: 10.1002/hep.1840140124. PMID 2066062